CLINICAL TRIAL: NCT00004248
Title: A Low Dose Schedule of Adriamycin and Protracted Infusion of Recombinant Interleukin-2: A Phase II Study of Immunotherapy in Unresectable Hepatocellular Carcinoma
Brief Title: Doxorubicin and Interleukin-2 in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Lawrance Liechman,MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000067494; RPCI-RP-9814
Record Dates: First submitted 2000-01-28; First posted 2004-03-31 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — aldesleukin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill liver cancer cells.

PURPOSE: Phase II trial to study the effectiveness of doxorubicin and interleukin- 2 in treating patients who have liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the immunological response to doxorubicin and protracted recombinant interleukin-2 in terms of alterations in hepatocellular carcinoma specific cytotoxic T cells detectable in peripheral blood in patients with unresectable hepatocellular carcinoma. II. Determine the toxicity of this treatment regimen in this patient population. III. Determine the tumor response to this regimen in terms of changes in alpha fetoprotein and tumor size measured by CT scan in these patients. IV. Determine the progression free survival and overall survival of this patient population treated with this regimen. V. Determine the correlation between immunological response, tumor response, progression free survival and overall survival in these patients.

OUTLINE: Patients receive doxorubicin IV over 3-5 minutes on day 1 and recombinant interleukin-2 (IL-2) IV continuously beginning on day 5 and continuing until day 57. Patients achieving partial or complete clinical response regardless of immunological response and patients with stable disease and an immunological response continue on IL-2 therapy continuously until day 92. Patients with stable disease and no immunological response receive an additional dose of doxorubicin on day 57 and then continue on IL-2 until day 92. Patients who are clinically eligible with progressive disease and an immunological response continue IL-2 therapy as above. Patients are followed at 2 weeks and then monthly thereafter.

PROJECTED ACCRUAL: A total of 24-30 patients will be accrued for this study within approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hepatocellular carcinoma OR Elevation of alpha fetoprotein (AFP) (greater than 400 ng/mL) in the presence of a space occupying lesion in the liver with known chronic liver disease Lesion must be easily biopsied Unresectable disease Bidimensionally measurable disease by radiography OR Evaluable disease with elevated AFP Okuda stage I disease Tumor size less than 50% of liver No ascites Albumin greater than 3 g/dL Bilirubin less than 2 mg/dL OR Okuda stage II disease Bilirubin as in stage I If ascites present, albumin must be greater than 3 g/dL

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Hemoglobin at least 9.0 g/dL Neutrophil count at least 1,500/mm3 Platelet count at least 80,000/mm3 Hepatic: See Disease Characteristics SGOT/SGPT no greater than 4 times upper limit of normal Any cause of underlying liver disease including hepatitis B or C allowed Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No poor cardiac function No myocardial infarction within the past 6 months No poorly controlled arrhythmia No congestive heart failure LVEF at least 45% by MUGA Other: No active hepatic encephalopathy No other active malignancies except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix HIV negative No immunodeficiency Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy, including interferon Chemotherapy: No prior systemic or intra arterial doxorubicin At least 6 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: At least 4 weeks since prior investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1999-07; Primary Completion 2000-06 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Albany Medical College
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States